CLINICAL TRIAL: NCT04566042
Title: A Novel ACT-based Video Game to Support Mental Health Through Embedded Learning: A Mixed-methods Feasibility Study Protocol
Brief Title: A Novel ACT-based Video Game
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, Darren Edwards, Senior Lecturer, Swansea University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Swansea U1
Record Dates: First submitted 2020-09-21; First posted 2020-09-28 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Depression; Anxiety; Stress, Emotional; Quality of Life; Psychological Flexibility; Social Connecedness
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT video game (Experimental)
  Interventions: Behavioral: Acceptance and commitment therapy video game

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy video game — The intervention is a videogame which teaches the participant about acceptance and commitment therapy.

SUMMARY:
A feasibility study to explore whether an acceptance and commitment therapy (ACT) can reduce mental health outcomes (stress, anxiety, depression) and increase psychological flexibility.

ELIGIBILITY:
Inclusion Criteria:

* Adults reporting some existing form of anxiety, depression or ongoing stress.
* Need ability to read and write English.
* Need internet access to play the videogame.

Exclusion Criteria:

* Those who are under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-07-31 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited for the study | 3 Weeks
  Feasibility outcome for recruitment.
Number of participants who completed all aspects of the study | 3 Weeks
  Feasibility outcome for retention of participants.
Reflexive thematic analysis themes | 3 Weeks; Immediate post intervention, and 3-week follow-up
  Acceptability of the intervention assessed through qualitative analysis of semi-structured interviews.

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale-21 (Depression subscale) | 3 Weeks; Baseline, immediate post intervention, and 3-week folllow-up
  Quantitative psychometric measure for depression. Score Range: Min=0, Max=21. Higher scores indicate higher depression.
Depression Anxiety Stress Scale-21 (Anxiety subscale) | 3 Weeks; Baseline, immediate post intervention, and 3-week folllow-up
  Quantitative psychometric measure for anxiety. Score Range: Min=0, Max=21. Higher scores indicate higher anxiety.
Depression Anxiety Stress Scale-21 (Stress subscale) | 3 Weeks; Baseline, immediate post intervention, and 3-week folllow-up
  Quantitative psychometric measure for stress. Score Range: Min=0, Max=21. Higher score indicate higher stress.
Acceptance and Action Questionnaire- second version | 3 Weeks; Baseline, immediate post intervention, and 3-week folllow-up
  Quantitative psychometric measure for psychological inflexibility. Score Range: Min=7, Max=49. Higher scores indicate higher psychological inflexibility.
Social Connectedness (adapted from Russell's (1996) University of California, Los Angeles Loneliness Scale) | 3 Weeks; Baseline, immediate post intervention, and 3-week folllow-up
  Quantitative psychometric measure of Social Connectedness. Score range: Min=2, Max=8. Higher scores indicate higher social connectedness.
Warwick-Edinburgh Mental Well-Being Scale | 3 Weeks; Baseline, immediate post intervention, and 3-week folllow-up
  Quantitative psychometric measure of mental well-being with a focus on positive aspects of mental health. Score Range: Min=14, Max=70. Higher scores indicate higher wellbeing.
EuroQol five dimensions (Mobility Subscale) | 3 Weeks; Baseline, immediate post intervention, and 3-week folllow-up
  Score Range: Min=1, Max=5. Higher scores indicate lower mobility.
EuroQol five dimensions (Self-care Subscale) | 3 Weeks; Baseline, immediate post intervention, and 3-week folllow-up
  Score Range: Min=1, Max=5. Higher scores indicate lower self-care.
EuroQol five dimensions (Usual Activities Subscale) | 3 Weeks; Baseline, immediate post intervention, and 3-week folllow-up
  Score Range: Min=1, Max=5. Higher scores indicate lower partaking in usual activities.
EuroQol five dimensions (Pain/Discomfort Subscale) | 3 Weeks; Baseline, immediate post intervention, and 3-week folllow-up
  Score Range: Min=1, Max=5. Higher scores indicate lower pain/discomfort.
EuroQol five dimensions (Anxiety/Depression Subscale) | 3 Weeks; Baseline, immediate post intervention, and 3-week folllow-up
  Score Range: Min=1, Max=5. Higher scores indicate lower anxiety/depression.
EuroQol five dimensions (Score to indicate how health is today) | 3 Weeks; Baseline, immediate post intervention, and 3-week folllow-up
  Score Range: Min=0, Max=100. Higher scores indicate higher health.

CONTACTS AND LOCATIONS:
Locations (1):
- Swansea University, Swansea, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gordon TC, Kemp AH, Edwards DJ. Mixed-methods feasibility outcomes for a novel ACT-based video game 'ACTing Minds' to support mental health. BMJ Open. 2024 Mar 29;14(3):e080972. doi: 10.1136/bmjopen-2023-080972. PMID 38553053
- [Derived] Edwards DJ, Kemp AH. A novel ACT-based video game to support mental health through embedded learning: a mixed-methods feasibility study protocol. BMJ Open. 2020 Nov 16;10(11):e041667. doi: 10.1136/bmjopen-2020-041667. PMID 33199427